CLINICAL TRIAL: NCT00508989
Title: Niacin Therapy to Improve Endothelial Function in Sickle Cell Disease
Brief Title: Niacin to Improve Blood Flow in People With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070196; 07-H-0196
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2015-12-24

CONDITIONS: Sickle Cell Disease
Keywords: Acetylcholine; Forearm Blood Flow; HDL; L-NMMA; Sickle Cell Anemia; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — omega-N-Methylarginine; Acetylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Niacin-ER; Drug: L-NMMA; Drug: Acetylcholine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niacin-ER — 500 mg daily for 4 weeks, 1000 mg daily for 4 weeks, and 1500 mg daily for 4 weeks
  Arms: 1
Drug: Placebo — 500 mg daily for 4 weeks, 1000 mg daily for 4 weeks, and 1500 mg daily for 4 weeks
  Arms: 2
Drug: L-NMMA
  Arms: 1
Drug: Acetylcholine
  Arms: 1

SUMMARY:
This study will determine whether niacin can improve blood flow in people with sickle cell disease, in which abnormal red blood cells interfere with blood flow to cause the disease symptoms. Niacin, a drug that has been used to increase HDL (good cholesterol) levels, improves blood flow in people without sickle cell disease. This study will see if it can do the same in people with the disease.

Patients with sickle cell disease between 18 and 65 years of age may be eligible for this study.

Candidates are screened with a medical history, physical examination, blood tests, echocardiogram and 6-minute walk test of exercise capacity.

Participants have the following baseline blood flow studies:

* Flow-mediated dilation (FMD): An ultrasound picture of the artery in the forearm is obtained. A blood pressure cuff is then placed on the upper arm and inflated for 5 minutes. After the pressure cuff is released, the ultrasound is repeated.
* Peripheral artery tonometry (PAT): A sensor is placed on the subject s finger. The sensor puts pressure on the finger and measures blood flow.
* Standard forearm blood flow test: Small tubes are placed in the artery of the forearm at the inside of the elbow. Saline is infused into one tube. Pressure cuffs are applied to the wrist and upper arm. A strain gauge (rubber band device) is placed around the forearm. When the cuffs are inflated, blood flows into the arm, stretching the strain gauge, and the flow measurement is recorded. Blood samples are collected from the tube in the artery to measure blood counts, proteins and other chemicals. At various times, small doses of the following drugs are administered through the tube in the vein:

  * Sodium nitroprusside causes blood vessels to dilate and increases blood flow to the heart.
  * Acetylcholine causes blood vessels to dilate and slows heart rate.
  * LNMMA decreases blood flow by blocking the production of nitric oxide.

Blood flow is measured after each dose of the different drugs. There are rest periods between injections of the different drugs. Pictures of the forearm are taken during the studies using an infrared camera and computer.

-Drug Treatment. Participants are assigned to take three 4-week courses of niacin or placebo. They return to the Clinical Center at the following intervals from the time they start the test drug for followup:

* Weeks 2, 6 and 10: Brief medical history, review of medication side effects and blood tests.
* Weeks 4 and 8: Physical examination, brief medical history, review of medication side effects and blood tests, repeat FMD and PAT blood flow studies and 6-minute walk test.
* Week 12: Same as weeks 4 and 8 plus standard blood flow studies and echocardiogram.

DETAILED DESCRIPTION:
Sickle cell disease is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15 percent of African-Americans are homozygous for sickle cell disease, and 8 percent have sickle cell trait. Hemoglobin S polymerization leads to red cell rigidity, microvascular obstruction, inflammation, and end-organ ischemic injury. Our published data indicate that up to 50 percent of sickle cell patients have vascular dysfunction due to impaired bioavailability of endogenous nitric oxide, due in large part to scavenging of nitric oxide by cell-free hemoglobin. We recently have completed studies that directly demonstrate endothelial dysfunction in patients with sickle cell disease, characterized by decreased ACh dependent vasorelaxation in forearm blood flow studies, distinct from the nitric oxide resistance above. Further, we have found in sickle cell patients a new association between low levels of apoA-I, pulmonary hypertension and endothelial dysfunction. Raising levels of HDL, and therefore apoA-1, could have the effect of ameliorating the endothelial dysfunction characteristic of sickle cell disease by affecting endothelium dependent vasorelaxation. Therapies directed at restoring HDL in these patients may be beneficial.

HDL is thought to promote vascular health in a variety of ways, some of which are unrelated to lipid transport. One of the best-known mechanisms relates to efflux of cholesterol from atherosclerotic plaque, yet HDL is thought to have several antithrombotic and anti-inflammatory effects. In vitro HDL attenuates formation of oxidized LDL and inhibits endothelial cell expression of inflammatory cell adhesion molecules. It is also thought to mediate NO production via stimulation of eNOS, thereby modulating endothelial function. In a study of subjects with atherosclerosis, low HDL levels correlated with impaired vasomotor relaxation via brachial artery FMD. Another study utilizing recombinant HDL cholesterol infused into brachial arteries of hypercholesterolemic men resulted in increased acetylcholine mediated blood flow that was inhibited by the infusion of L-NAME, an eNOS inhibitor, suggesting that HDL increased blood flow via an eNOS dependent mechanism. This may have implications not only for subjects with atherosclerosis, but also for those with sickle cell disease and endothelial dysfunction.

We propose that niacin therapy could improve vascular reactivity in response to acetylcholine. Several options for increasing HDL levels have been previously utilized in forearm flow studies using venous occlusion plethysmography or flow-mediated dilation. Reconstituted HDL (rHDL), apoA-1 mimetics and niacin therapy were all shown to improve endothelial dysfunction, and proved safe and effective.

This trial will aim to 1) establish the effects of niacin treatment on raising HDL levels in subjects with sickle cell disease, 2) investigate whether niacin treatment would result in improvement of endothelial-dependent relaxation via venous occlusion plethysmography, and 3) compare the efficacy of peripheral arterial tonometry measurements to venous occlusion plethysmography and flow-mediated dilation as indicators of vascular dysfunction.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males or females 18 to 65 years of age.
* Diagnosis of sickle cell disease (electrophoretic or HPLC documentation of hemoglobin S only phenotype is required).
* Hemoglobin greater than 5.5 grams per deciliter
* Absolute reticulocyte count greater than 95,000 microliters if hemoglobin is less than 9.0 grams per deciliter.
* An apoA-1 level lower than 99 milligrams per deciliter (median value among sickle cell subjects), or HDL-C level below 39 milligrams per deciliter (median value amongst our sickle cell cohort).

EXCLUSION CRITERIA:

* Acute pain crisis requiring intravenous analgesics within the last week.
* Current pregnancy or lactation.
* Hemoglobin SC disease, or hemoglobin A greater than 20%
* Conditions that may independently affect endothelial function:

  1. Diabetes mellitus
  2. Cigarette smoking within one month
  3. Uncontrolled hypertension
* Serum creatinine greater than 2.0 milligram per deciliter
* Serum alanine aminotransferase (ALT) greater than 3 times the upper limit of normal. (AST elevation will not be used as an exclusion criterion, since this is elevated in normal sickle cell subjects due to red cell lysis, even without liver injury)
* Uric acid level greater than 8 or history of gout
* History of GI bleeding within the past 6 months
* Active peptic ulcer disease
* Hemoglobin less than or equal to 5.5 grams per deciliter; however, subjects may return for evaluation at a later date.
* No aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) for 1 week prior to forearm blood flow assessment and no caffeine the day of each forearm blood flow study. Subjects on opiates or acetaminophen will not be excluded.
* Subjects taking sildenafil, vardenafil, tadalafil, L-arginine, fibrates (e.g., clofibrate, gemfibrozil, or fenofribrate) or inhaled nitric oxide within the last week will be excluded from the study.
* Subjects taking any statin drug (e.g., fluvastatin, lovastatin, pravastatin, simvastatin, rosuvastatin) within the last four weeks will be excluded from the study.
* Subjects taking prostaglandins such as epoprostenol or treprostinil will be excluded from the study.
* Subjects with significant cardiac disease and/or known peripheral Arterial disease.
* Subjects with significant hypotension.
* Women who do not use birth control while participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07-24; Primary Completion 2010-12-31 (Actual); Study Completion 2015-12-24 (Actual)

PRIMARY OUTCOMES:
The Effect of niacin-ER on endothelial dysfunction in the sickle cell. | 12 weeks

SECONDARY OUTCOMES:
Effect of niacin therapy on HDL and apo A-I levels in subjects with sickle cell disease. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Howard University Hospital, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Barter PJ, Nicholls S, Rye KA, Anantharamaiah GM, Navab M, Fogelman AM. Antiinflammatory properties of HDL. Circ Res. 2004 Oct 15;95(8):764-72. doi: 10.1161/01.RES.0000146094.59640.13. PMID 15486323
- [Background] Kwiterovich PO Jr. The antiatherogenic role of high-density lipoprotein cholesterol. Am J Cardiol. 1998 Nov 5;82(9A):13Q-21Q. doi: 10.1016/s0002-9149(98)00808-x. PMID 9819099
- [Background] Viswambharan H, Ming XF, Zhu S, Hubsch A, Lerch P, Vergeres G, Rusconi S, Yang Z. Reconstituted high-density lipoprotein inhibits thrombin-induced endothelial tissue factor expression through inhibition of RhoA and stimulation of phosphatidylinositol 3-kinase but not Akt/endothelial nitric oxide synthase. Circ Res. 2004 Apr 16;94(7):918-25. doi: 10.1161/01.RES.0000124302.20396.B7. Epub 2004 Feb 26. PMID 14988229